CLINICAL TRIAL: NCT06816160
Title: Tru-cut Biopsy in Tumor Characterisation
Acronym: TRUTH
Status: Recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Renata Poncová, Principal Investigator, General University Hospital, Prague
Other Study IDs: 10/23 Grant GIP
Record Dates: First submitted 2024-03-02; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Tumor
Keywords: tumor; biopsy; tru-cut; core-cut; cancer; pelvic tumor
MeSH Terms: conditions — Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy from tumor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: tru-cut biopsy — needle biopsy from the tumor
  Other Names: core-cut biopsy

SUMMARY:
Tru-cut biopsy (TCB) is a minimally invasive method to get an adequate sample from the lesion in order to tailor the appropriate management avoiding unnecessary surgery. The aim of our trial is to evaluate the adequacy, accuracy and safety of the method related to the final histology as reference standard.

DETAILED DESCRIPTION:
The primary endpoint is represented by the assessment of adequacy, accuracy and safety of the procedure in prospective settings. The secondary endpoint is to evaluate feasibility of immunohistochemistry (IHC), next generation sequencing (NGS) and tumor immunology in obtained samples by TCB and to assess the alterations of these tumor characteristics in relation to the treatment. The additional endpoint includes the effect of several variables (e.g. tumor origin, size of the tumor, presence of ascites, body mass index (BMI), biopsy site, biopsy approach - transvaginal, transrectal vs. transabdominal, status of the disease - the first diagnosis, the first and other recurrence or progression and previous treatment modality - chemotherapy, anti-angiogenic therapy, PARP inhibitor therapy, hormonal therapy, radiotherapy) on the outcome of the procedure (adequacy, accuracy and safety).

All patients indicated for tru-cut biopsy (including advanced stages of ovarian, endometrial or cervical cancers) in Gynecologic Oncology Center of the General University Hospital from February 2024 to January 2026 will be recruited. Furthermore, all patients with suspicious recurrence or progression of already known gynecologic malignancy based on the imaging methods will be recruited. The duration of recruitment is 3 years, and we expect 250 patients enrolled into the trial. Data will be assessed in relation to the patient characteristics, tumor/lesion characteristics, procedure specifications, histopathological characteristics and IHC/NGS/immunological characteristics, consequent biopsy/surgery and final histopathological results. All adverse events will be recorded. Moreover, patient related outcomes will be recorded within 72 hours after the procedure.

This prospective study could support our hypothesis that TCB is feasible and safe procedure with high adequacy and accuracy rate. It enables to get appropriate outcomes of IHC, NGS and immunology preoperatively. We expect that TCB is applicable and efficient in majority of recurrences/disease progressions, so it can be considered suitable technique for de novo biopsy. It can help us show the alterations of tumor characteristics after the previous treatment and can be used to select appropriate targeted therapy.

ELIGIBILITY:
Inclusion Criteria: Presence of a pelvic/abdominal lesion with suspicion of malignancy:

1. new diagnosis of a presumed gynecologic tumor
2. suspicious recurrence or progression of a known gynecologic malignancy
3. pelvic/abdominal spread or recurrence of a non-gynecologic tumor (primary tumor or metastasis)
4. pelvic/abdominal spread of a tumor of unknown origin 2. Age ≥18 years 3. Eastern Cooperative Oncology Group (ECOG) performance status grade <3 4. Not pregnant 5. Signed informed consent form

Exclusion Criteria:

1. Considered by the investigator to be unsuitable for any treatment
2. Early stage disease
3. Age <18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women
Study Population: Women with abdominopelvic tumor
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The adequacy of samples obtained by TCB for histopathological examination (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  1. The adequacy means the ability to determine the type of tumor (in %)

SECONDARY OUTCOMES:
The adequacy of samples obtained by TCB for next-generation sequencing examination (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  2. Adequacy of samples obtained by TCB for next-generation sequencing examination (in %) Adequacy is defined as the ability to determine the complex classification of the tumor.
The adequacy of samples obtained by TCB for immunohistochemistry examination (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  3. Adequacy of samples obtained by TCB for immunohistochemistry examination (in %) Adequacy is defined as the ability to determine the complex classification of the tumor.
The adequacy of samples obtained by TCB for immunologic examination (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  4. Adequacy of samples obtained by TCB for immunologic examination (in %) Adequacy is defined as the ability to determine the complex classification of the tumor.

OTHER OUTCOMES:
1. To evaluate which factors affect the primary and secondary endpoints 2. To evaluate the overall safety of TCB (in %) 3. To evaluate the overall accuracy of TCB for complex classification of pelvic and abdominal tumors (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  5. Evaluation of factors affecting the primary and secondary endpoints
  Includes tumor origin, size, presence of ascites, BMI, biopsy site, biopsy approach, disease status, and previous treatment modalities.
Overall safety of TCB (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  6. Overall safety of TCB (in %)
Overall accuracy of TCB for complex classification of pelvic and abdominal tumors (in %) | First data 31st of June 2025, definitive data 31st of January 2026
  7. Overall accuracy of TCB for complex classification of pelvic and abdominal tumors (in %)

CONTACTS AND LOCATIONS:
Overall Officials: David Cibula, prof., Study Chair — Department of Gynecology, Obstetrics and Neonatology
Locations (1):
- Department of Gynecology, Obstetrics and Neonatology of First Faculty of Medicine and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Registration of subjects into the database using the REDCap (Research Electronic Data Capture, www.projectredcap.org) electronic data capture tool.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1.2.2024 - 31.1.2026
Access Criteria: Study participation
URL: http://redcap.lf1.cuni.cz/

DOCUMENTS (2):
  • Study Protocol (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06816160/Prot_000.pdf
  • Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT06816160/ICF_001.pdf